CLINICAL TRIAL: NCT00270829
Title: Renal Effects of Intrarenal Nesiritide
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding not available
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Steve Gottlieb, Professor o Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-26854
Record Dates: First submitted 2005-12-23; First posted 2005-12-28 (Estimated); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Heart Failure, Congestive
Keywords: renal function
MeSH Terms: conditions — Heart Failure | interventions — Natriuretic Peptide, Brain

ARMS (2):
- 1 (Experimental): Nesiritide given intrarenally
  Interventions: Drug: nesiritide
- 2 (No Intervention): No intrarenal drug administration

INTERVENTIONS:
Drug: nesiritide — Drug given intrarenally or placebo
  Arms: 1

SUMMARY:
The impact of nesiritide in CHF is unclear, but it is possible that systemic vasodilation leads to adverse consequences even if the direct renal effects are positive. Therefore, this study will look at the effects of direct intrarenal administration of nesiritide on GFR and RPF.

DETAILED DESCRIPTION:
We will perform an open-label, parallel arm, controlled study of intrarenal nesiritide in 26 patients hospitalized with CHF. Patients will be admitted for CHF exacerbation and randomly but equally divided into treatment and placebo groups. Both arms will receive diuretics on admission as dictated by clinical need. They will then have an 8-hour diuretic-free period (overnight). Each arm will then have renal parameters (GFR, RPF, urine output, urinary sodium excretion) assessed using PAH and iothalamate. These parameters will be measured prior to administration of drug during period 1. Randomization will be performed via an interactive computerized call in program following completion of screening procedures and once patient has given informed consent.

At time 0, treatment patients will be taken to the cardiac catheterization lab for placement of the Benephit Infusion System (Flow Medica). Placement involves femoral artery cannulation and introduction of a bifurcated infusion catheter into the arterial system to a destination at the level of renal arteries. This will be done under fluoroscopic guidance.

When placement of catheter is completed, period 2 will begin with initiation of Study Drug infusion (IR nesiritide or IV D5W). Nesiritide will be diluted according to its labeled instructions in D5W to a final dilution of 6 mcg/mL. Placebo patients will receive IV D5W as a bolus and a continuous infusion of D5W at volumes equal to what they would have gotten had they been randomized to nesiritide.

Intra-renal (IR) infusion of nesiritide will be given as a 2ug/kg bolus followed by an infusion of 0.01 mg/kg/min through the intrarenal catheter. The nesiritide infusion will continue for 6 hours.

Period 3 begins at the 3-hour mark, at which time, both the placebo and treatment groups will be treated with boluses of intravenous furosemide. Both treatment arms will receive furosemide at this time. Blood drawn at 3 and 6 hours and urine collected between 3 and 6 hours will be used to determine GFR, RPF, Na excretion and urine output.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for worsening CHF and volume overload
* Creatinine increased by greater than or equal to 0.2 and greater than or equal to 10% above baseline at study initiation
* Age greater than or equal to 18 years
* NHYA class II-IV at the time of initiation in the study
* EF less than or equal to 40%
* Signed Informed Consent

Exclusion Criteria:

* Current or anticipated need for dialysis during the study period
* Systolic blood pressure less than or equal to 90 mmHg
* Calculated CrCL based on Cockcroft-Gault less than or equal to 15 cc/min
* Hypersensitivity to nesiritide
* Cardiogenic shock
* Clinically significant aortic or mitral stenosis
* Contraindication to vasodilator treatment
* Inability to withstand 11-15 hours without diuretics
* Suspected renal deterioration due to causes unrelated to CHF such as radiocontrast administration, NSAID use
* Receipt of dose of NSAID within 12 hours of study drug initiation
* Use of radiocontrast media within 7 days of study drug initiation (other than the small amount of IV contrast that will be needed to place intrarenal catheter to the level of the renal artery)
* Use of nephrotoxic drugs such as aminoglycosides or cisplatinum within 7 days of study initiation
* Use of sildenafil or other PDE5 inhibitors within 24 hours of study drug initiation
* Diseases of weak collagen (i.e. Marfans)
* Aortic or renal aneurysm
* Significant calcification in the region of the renal ostia, or any other condition that would, in the opinion of the investigator, increase risk of placement of an intravascular sheath and catheter.
* Known bleeding diathesis
* Solitary kidney or solitary functioning kidney
* Known uncorrected renal artery stenosis greater than 50% in either renal artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
GFR | hours

SECONDARY OUTCOMES:
Urine output | hours
RPF | hours
sodium excretion | hours

CONTACTS AND LOCATIONS:
Overall Officials: Stephen S Gottlieb, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland, Baltimore, Maryland, United States